CLINICAL TRIAL: NCT07126223
Title: The Effect of Hot Water Foot Bath on Pain and Gas Release After Laparoscopic Cholecystectomy: A Randomised Controlled Trial
Brief Title: Hot Water Foot Bath for Pain and Gas Relief After Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cansu Mert (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, Cansu Mert, Lecturer, Fenerbahce University
Organization: Fenerbahce University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 103.2024fbu
Record Dates: First submitted 2025-07-23; First posted 2025-08-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Pain; Gastrointestinal Motility; Postoperative Recovery; Nursing Interventions
Keywords: foot bath; gas release; pain management; complementary therapy; nursing; cholesistectomy
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: the intervention group receiving a hot foot bath and the control group receiving standard postoperative care. Both groups will be monitored concurrently without crossover throughout the study.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor responsible for recording postoperative pain levels and time to first flatus will be blinded to group allocation in order to reduce measurement bias. Participants and care providers cannot be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot water foot bath group (Experimental): Participants in this group will receive a 20-minute hot foot bath using a device with fixed temperature control (41°C), anti-slip base, timer, and vibration massage features. The intervention will be conducted 3 hours after postoperative transfer to the ward, once the patient is clinically stable. The room temperature will be maintained between 22°C and 25°C throughout the intervention. Participants will sit in a chair and immerse their feet in 41°C water for 20 minutes. Afterward, their feet will be wrapped in a towel for 10 minutes to retain heat. Pain levels (NRS) will be assessed immediately before the intervention, and again at 1 and 2 hours post-intervention (corresponding to 4h30 and 5h30 post-surgery). Time to first flatus will also be tracked using a monitoring form filled by patients or caregivers.
  Interventions: Behavioral: Hot water foot bath
- Standard postoperative care group (No Intervention): Participants in this group will receive standard postoperative care without any foot bath intervention. Pain levels (NRS) will be evaluated at 3h30, 4h30, and 5h30 after surgery. Room temperature will be maintained between 22°C and 25°C. First gas passage time will be tracked using a monitoring form completed by the patient or caregiver.

INTERVENTIONS:
Behavioral: Hot water foot bath — A 20-minute hot foot bath therapy using a specially designed foot spa device (41°C) applied in the early postoperative period. Follow-up includes pain evaluation via Numeric Rating Scale (NRS) and monitoring of first flatus time.
  Arms: Hot water foot bath group

SUMMARY:
This study investigates the effects of a hot foot bath on postoperative pain and time to first gas release in patients undergoing laparoscopic cholecystectomy. The intervention is a non-pharmacological supportive method applied during the early postoperative period. Participants will be randomly assigned to either intervention or control groups. No FDA-regulated drug or device is involved.

DETAILED DESCRIPTION:
This randomised controlled clinical trial aims to evaluate the effects of hot foot bath therapy on postoperative pain and time to first flatus in patients undergoing laparoscopic cholecystectomy. The hot water foot bath is a non-pharmacological, supportive intervention to be administered at 3 hours postoperatively after patients have regained consciousness and are clinically stable.

Participants will be randomly divided into two groups: the intervention group will receive a 20-minute foot bath at a water temperature of 41°C, while the control group will receive standard postoperative care without a foot bath. The primary outcomes include pain level assessed using the Numerical Rating Scale (NRS) and time to first flatus recorded in hours postoperatively.

In addition to these primary outcomes, the study will also collect data through a two-part questionnaire. The first part will include questions regarding the sociodemographic and medical history of the patients, such as age, gender, marital status, education level, income level, presence of chronic diseases, previous surgical history, preoperative bowel movement frequency and duration of surgery. The second part focuses on indicators of postoperative recovery, including time to surgery, time to postoperative ward arrival, time to first oral intake, time to first mobilisation, total mobilisation time in the first 8 hours, time to first gas passage and type of analgesic administered.

This study does not involve any drug or device regulated by the U.S. Food and Drug Administration (FDA). Ethical approval was obtained from the Fenerbahçe University Non-Interventional Research Ethics Committee. Institutional permission was also granted in writing by Istanbul University-Cerrahpaşa Faculty of Medicine Hospital, where the clinical study will be conducted. No funding was received from Fenerbahçe University or any other organization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing elective laparoscopic cholecystectomy
* Received the same preoperative gastrointestinal preparation protocol
* Received the same postoperative analgesia protocol
* Numeric Rating Scale (NRS) pain score of 3 or higher at the 3rd postoperative hour
* Voluntarily agreed to participate and signed the informed consent form
* Classified as ASA I or ASA II according to the American Society of Anesthesiologists (ASA)

Exclusion Criteria:

* Undergoing emergency cholecystectomy or open surgery (laparotomy)
* Presence of open wounds, infections, circulatory disorders, or lesions in the feet (hot foot bath area)
* Use of patient-controlled analgesia (PCA) in the early postoperative period
* Any condition that impairs verbal communication
* History of inflammatory bowel disease (due to potential influence on bowel motility)
* Use of medications or probiotic agents affecting bowel motility in the pre- or postoperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity at 3 hours after transfer to the ward (pre-intervention baseline) | 3 hours after transfer to the ward
  Pain intensity will be assessed using the 11-point Numeric Rating Scale (0 = no pain, 10 = worst pain imaginable). Higher scores indicate worse outcomes.
Postoperative pain intensity at 1 hour after the intervention | 1 hour after the intervention
  Pain intensity will be assessed using the 11-point Numeric Rating Scale (0 = no pain, 10 = worst pain imaginable). Higher scores indicate worse outcomes.
Postoperative pain intensity at 2 hours after the intervention | 2 hours after the intervention
  Pain intensity will be assessed using the 11-point Numeric Rating Scale (0 = no pain, 10 = worst pain imaginable). Higher scores indicate worse outcomes.
Time to first postoperative gas release | Up to 72 hours postoperatively
  The time (in hours) from the end of surgery to the first postoperative gas release will be recorded. Patients or caregivers will use a monitoring form to document the exact time of gas passage, which will be confirmed by the research team during routine postoperative follow-up.

SECONDARY OUTCOMES:
Total dose of analgesic medication used within the first 24 hours postoperatively | 0-24 hours after surgery
  Total amount of analgesics (e.g., paracetamol, NSAIDs, opioids) administered and/or requested will be recorded from medical records.
Age (years) | Baseline (upon study entry)
  Participant age will be recorded from medical records in years.
Sex | Baseline (upon study entry)
  Participant sex (male/female) will be recorded.
Body Mass Index (BMI) | Baseline (upon study entry)
  BMI will be calculated based on weight (kg) and height (m) and recorded as kg/m².
ASA Physical Status Classification | Baseline (upon study entry)
  ASA physical status classification will be noted from the preoperative anesthesia evaluation
Type of anesthesia | Baseline (upon study entry)
  Type of anesthesia administered (general/regional) will be recorded.
Surgical duration | From skin incision to skin closure
  Duration of the surgical procedure (in minutes) will be recorded.
Comorbidities | Baseline (upon study entry)
  Pre-existing comorbid conditions will be documented using structured data form.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study does not include prior approval from the ethics committee or institutional policies for data sharing. Additionally, no data sharing was planned in the informed consent obtained from participants.